CLINICAL TRIAL: NCT01425567
Title: Compassionate Use of an Intravenous Lipid Emulsion Comprised of Fish Oil in the Treatment of Parenteral Nutrition Induced Liver Injury in Children
Brief Title: Compassionate Use of IV Fish Oil for Parenteral Nutrition (PN) Liver Injury
Acronym: Omegaven
Status: Approved for marketing | Type: Expanded Access
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC2011-0211T
Record Dates: First submitted 2011-08-03; First posted 2011-08-30 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Liver Disease
Keywords: cholestasis; parenteral nutrition
MeSH Terms: conditions — Liver Diseases; Cholestasis; Hyperphagia | interventions — fish oil triglycerides

INTERVENTIONS:
Drug: Intravenous Lipid Emulsion Comprised of Fish Oil — IV lipid provided for parenteral nutrition when enteral feeds are not tolerated due to intestinal disease
  Other Names: Omegaven

SUMMARY:
To establish a process by which critically ill infants with parenteral nutrition-associated liver disease can receive a fish oil-based intravenous lipid emulsion (Omegaven®) for compassionate use when no satisfactory alternative treatments are available.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria (having a direct bilirubin ≥4.0 mg/dL) and are consented will be discontinued from standard soybean-based lipid emulsion and started on Omegaven®. Omegaven® will be infused continuously via either a peripheral or central catheter at a dose of 1 gm/kg/day along with parenteral nutrition (PN).

ELIGIBILITY:
Inclusion Criteria :

- >14 days <24 months* Anatomic short gut (< 50 % bowel removed) with total bilirubin > or = 4 mg/dL Or severe dysmotility of gut reflecting non functional gut with total bilirubin > or = 4 mg/dL Receiving at least 60 % calories by intravenous infusion Requires IV nutrition an additional 28 days * Patients with direct bilirubin > or = 6 mg/dL who do not meet criteria above but meet criteria with * If infants qualify for high risk ARM (gastroschisis, ileal atresia, <750 grams and stage III NEC) d bilirubin >1 mg/dL but less than 4 mg/dL.

Exclusion Criteria:

Congenital lethal condition (e.g. Trisomy 13) Clinically severe bleeding Evidence of viral hepatitis or primary liver disease as etiology of their cholestasis Other health problems such as survival extremely unlikely even if cholestasis improves Known allergies to eggs or shellfish

Ages: 14 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Blanco, MD, Principal Investigator — University of Texas
Locations (1):
- University Health System, San Antonio, Texas, United States

REFERENCES:
- [Derived] Sorrell M, Moreira A, Green K, Jacob R, Tragus R, Keller L, Quinn A, McCurnin D, Gong A, El Sakka A, Mittal N, Blanco C. Favorable Outcomes of Preterm Infants With Parenteral Nutrition-associated Liver Disease Treated With Intravenous Fish Oil-based Lipid Emulsion. J Pediatr Gastroenterol Nutr. 2017 May;64(5):783-788. doi: 10.1097/MPG.0000000000001397. PMID 28437326